CLINICAL TRIAL: NCT02623790
Title: Study of the Impact of Cheese Matrix on Postprandial Lipemia: a Clinical Study
Acronym: FROMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Couture, MD, PhD, FRCP, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Fromage-INAF
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Healthy
MeSH Terms: interventions — Butter

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test meal (butter) (Experimental): Subjects will eat one test meal containing 33g of lipids from butter (percent of total caloric intake: 15.0% from proteins; 53.0% from carbohydrates; 32.0% from fat).
  Interventions: Other: Test meal (butter)
- Test meal (cheddar cheese) (Experimental): Subjects will eat one test meal containing 33g of lipids from cheddar cheese (percent of total caloric intake: 15.0% from proteins; 53.0% from carbohydrates; 32.0% from fat).
  Interventions: Other: Test meal (cheddar cheese)
- Test meal (cream cheese) (Experimental): Subjects will eat one test meal containing 33g of lipids from cream cheese (percent of total caloric intake: 15.0% from proteins; 53.0% from carbohydrates; 32.0% from fat).
  Interventions: Other: Test meal (cream cheese)

INTERVENTIONS:
Other: Test meal (butter) — Subjects will eat one meal test containing 33g of lipids from butter (percent of total caloric intake: 15.0% from proteins; 53.0% from carbohydrates; 32.0% from fat).
  Arms: Test meal (butter)
Other: Test meal (cheddar cheese) — Subjects will eat one meal test containing 33g of lipids from cheddar cheese (percent of total caloric intake: 15.0% from proteins; 53.0% from carbohydrates; 32.0% from fat).
  Arms: Test meal (cheddar cheese)
Other: Test meal (cream cheese) — Subjects will eat one meal test containing 33g of lipids from cream cheese (percent of total caloric intake: 15.0% from proteins; 53.0% from carbohydrates; 32.0% from fat).
  Arms: Test meal (cream cheese)

SUMMARY:
Dairy products consumption is widely recommended in a healthy diet not only for bone growth and maintenance, but also as a protein, calcium and magnesium sources for an adequate diet. However, dairy products are a major dietary source of saturated fat that is associated with increased risk of coronary heart disease. ln this context, dietary guidelines still advocate a restriction in dietary saturated fat for optimal heart health. Nevertheless, the association between saturated fat and the risk of heart disease remains highly controversial within the scientific community. There is also emerging evidence that the impact of dietary saturated fat will be significantly influenced by the food matrix through which it is provided. Recent studies indicate that cheese could have a major influence on intestinal fat absorption and the magnitude of the after meal release of fat in blood circulation. This is of interest because substantial evidence exists indicating that elevated levels of the after meal fat levels are associated with increased cardiovascular risk. Therefore, the improvement of the after meal fat levels produced by cheese consumption could well be part of novel therapeutic approaches contributing to improve cardiovascular risk.

The general objective of the proposed research is to investigate how cheese consumption affects the after meal release of fat in blood circulation in healthy subjects. Our hypothesis is that, compared to butter, cheese consumption will have a beneficial impact on the after meal fat levels in healthy subjects. Favourable results from the proposed study will provide novel and much warranted evidence on the importance of considering changes in the after meal fat levels, not only bad cholesterol, as part of the on-going saturated fat-heart disease debate and that cheese should indeed be part of a healthy diet.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years (men and women)

Exclusion Criteria:

* Smokers (more than 1 cigarette/d)
* Body weight variation more than 10% during the last 6 months prior to the study baseline
* BMI more than 35 kg/m2
* Previous history of cardiovascular disease
* Subjects with type 2 diabetes
* Subjects with monogenic dyslipidemia
* Subjects taking anti-inflammatory drugs
* Subjects with endocrine or gastrointestinal disease
* Allergy/intolerance to dairy
* Clinical use of vitamin D and calcium supplements
* Vegetarians
* Subjects who are in situation or have a condition that, in the opinion of the investigators, may interfere with optimal participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in triglyceride concentrations 4h following the test meals ingestion | At week 0, week 2 and week 4 (at the end of the three test meals).

SECONDARY OUTCOMES:
Change in triglyceride concentrations (area under the curve) following the test meals ingestion | At week 0, week 2 and week 4 (at the end of the three test meals).
Change in free fatty acids concentrations (area under the curve) following the test meals ingestion | At week 0, week 2 and week 4 (at the end of the three test meals).
Change in apolipoprotein B48 concentrations (area under the curve) following the test meals ingestion | At week 0, week 2 and week 4 (at the end of the three test meals).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, PhD, FRCP, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drouin-Chartier JP, Tremblay AJ, Maltais-Giguere J, Charest A, Guinot L, Rioux LE, Labrie S, Britten M, Lamarche B, Turgeon SL, Couture P. Differential impact of the cheese matrix on the postprandial lipid response: a randomized, crossover, controlled trial. Am J Clin Nutr. 2017 Dec;106(6):1358-1365. doi: 10.3945/ajcn.117.165027. Epub 2017 Oct 4. PMID 28978543